CLINICAL TRIAL: NCT00381446
Title: Evaluation of Corneal Staining With Market Contact Lens/Solution Combinations
Brief Title: Evaluation of Corneal Staining With Various Contact Lens/Solution Combinations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Andrasko, Gary, OD, LLC (Individual)
Collaborators: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: MS005
Record Dates: First submitted 2006-09-25; First posted 2006-09-27 (Estimated); Last update posted 2007-09-27 (Estimated); Status verified 2007-09

CONDITIONS: Corneal Epithelial Disruption; Corneal Staining
Keywords: corneal staining; contact lens care; multipurpose solution

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Device: Marketed contact lens care products

SUMMARY:
The purpose of this study is to quantify the amount of corneal staining observed with various marketed contact lens/multipurpose solution combinations. The hypothesis is that there are measurable differences in the amount of corneal staining between the various combinations.

DETAILED DESCRIPTION:
A series of clinical studies is being conducted at one research site using a double-masked, randomized cross-over design. Each study consists of asymptomatic daily wear soft contact lens wearers observed at baseline and at two and four hours post lens insertion. Corneal staining is being assessed using sodium fluorescein, a cobalt filter and a yellow filter. Subjective comfort assessments are obtained at each visit.

ELIGIBILITY:
Inclusion Criteria:

* currently wearing soft contact lenses daily wear for at least 2 weeks prior to study
* correct visual acuity of 20/30 or better each eye

Exclusion Criteria:

* history of hypersensitivity to any components of solution being tested
* any ocular condition prohibiting contact lens wear
* excessive baseline staining as defined in protocol
* use of topical or OTC ocular medications during the study
* seasonal allergies with significant effect on contact lens wear

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2005-07; Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
Area of Corneal Staining

SECONDARY OUTCOMES:
Type (severity) of Corneal Staining

CONTACTS AND LOCATIONS:
Overall Officials: Gary J. Andrasko, OD, MS, Principal Investigator
Locations (1):
- Dr. Richard Erdey office, Columbus, Ohio, United States